CLINICAL TRIAL: NCT04966013
Title: A Phase II, Randomized, Sham Controlled Dose Finding Study of the RD-X19 Treatment Device in Individuals With Mild to Moderate COVID-19
Brief Title: Evaluation of the RD-X19 Treatment Device in Individuals With Mild to Moderate COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmitBio Inc. (Industry)
Responsible Party: Sponsor
Organization: KNOWBio Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB-P20-01
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Volunteers meeting all inclusion criteria and none of the exclusion criteria will be randomized to the RD-X19 treatment arm or the sham treatment arm within each cohort in a 2:1 ratio according to a fixed schedule via a permuted block design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- RD-X19 Device, Dose A (Active Comparator): RD-X19. Investigational device that delivers 24 J/cm2 of electromagnetic energy to the oropharynx.
  Interventions: Device: RD-X19
- RD-X19 Device, Dose B (Active Comparator): RD-X19. Investigational device that delivers 32 J/cm2 of electromagnetic energy to the oropharynx.
  Interventions: Device: RD-X19
- Sham Device (Sham Comparator): Investigational device that uses safe electromagnetic energy to target the oropharynx but at energy levels with a lower inactivation potential against SARS-CoV-2 in vitro.
  Interventions: Device: Sham

INTERVENTIONS:
Device: RD-X19 — Investigational device that uses safe electromagnetic energy to target the oropharynx.
  Arms: RD-X19 Device, Dose A; RD-X19 Device, Dose B
Device: Sham — Investigational device that uses safe electromagnetic energy to target the oropharynx but at energy levels with a lower inactivation potential against SARS-CoV-2 in vitro..
  Arms: Sham Device

SUMMARY:
This is a randomized, sham controlled, dose finding study of the EmitBio RD-X19 device in individuals with symptomatic COVID-19 in the outpatient setting.

DETAILED DESCRIPTION:
This is a randomized, sham controlled, dose finding study of the EmitBio RD-X19 device in individuals with symptomatic COVID-19 in the outpatient setting. Study subjects will self-administer treatment twice daily for 7 days with a one-week follow-up period at Day 14 (+/- 2 days) and will not be aware of which treatment group to which they have been randomized. Clinical outcomes will be assessed via patient reported outcomes (questionnaire and diary cards) and virologic outcomes will be assessed post baseline on Days 3, 5, 8, and 14 via biospecimen collection.

The primary goal of the study is to evaluate multiple doses of the RD-X19 treatment device and establish evidence for safety and efficacy for each of the RD-X19 doses compared to sham in SARS-CoV-2 infected individuals with outpatient COVID-19. The primary efficacy outcome is time to sustained symptom resolution. Other clinical and microbiological outcomes will also be assessed.

Safety and tolerability (local reactogenicity) will be assessed actively and study subject diary card data recorded at each clinic visit by review of potential treatment emergent adverse events (TEAEs) and targeted oral and physical examinations. Volunteers will be instructed to contact designated clinical trial staff for AEs of a medically-urgent nature as soon as is practically possible and to seek immediate medical care, if needed. Study subjects who experience progression of disease to a grade 3 severity score (e.g SpO2 ≤ 93%, or respiratory rate ≥30/ minute on room air) will be instructed to urgently seek medical care at their nearest Urgent Care or Emergency Department. Study subjects who progress to severe acute respiratory distress syndrome with substantial risk for mortality without immediate medical intervention will be referred directly by site staff to their closest hospital. All study subjects who are hospitalized will be tracked to assess time to hospital discharge or death; the time and date of these events will be captured as part of the trial data.

Metabolic, liver, kidney and hematological laboratory evaluations will be performed at baseline and at Day 14 or early termination (and potentially during unscheduled) clinic visits. Methemoglobin assessments will be performed at baseline and Day 14.

ELIGIBILITY:
Inclusion Criteria

1. Positive for SARS-CoV-2 as detected using an FDA authorized SARS-CoV-2 antigen test at or within 24 hours of the screening visit.
2. COVID-19 signs and symptoms within 72 hours from symptom onset, including at least two moderate* or greater symptoms from: cough, sore throat, nasal congestion, headache, unexplained chills and/or sweats, myalgia, fatigue, nausea (with or without vomiting).

   o Alternatively, subjects with the presence of at least one moderate symptom and either a) a fever with an oral temperature of at least 100.5° F or b) shortness of breath/difficulty breathing on exertion (e.g., walking, going up and down stairs) are also eligible for enrollment.
3. BMI <40
4. Provides written informed consent prior to initiation of any study procedures.
5. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
6. Agrees to the collection of saliva, nasopharyngeal, and venous blood specimens per protocol.
7. Males or females, 18 to 65 years of age, inclusive.
8. No uncontrolled disease process(es) based on patient reported medical history (chronic or acute), other than direct COVID-19 signs and symptoms.
9. No physical or mental conditions or attributes at the time of screening, which in the opinion of the PI, will prevent full adherence to, and completion of, the protocol.

   * Symptom scoring is independent from the classification of COVID-19 disease severity at baseline. Guidance to study subjects for grading of signs and symptoms will be based on definitions used for the grading of TEAEs:

     * None (Grade 0): Not present
     * Mild (Grade 1): Symptoms that are usually transient and may require only minimal or no palliative or specific therapeutic intervention and generally do not interfere with the subject's usual activities of daily living.
     * Moderate (Grade 2): Symptoms that are usually alleviated with palliative or specific therapeutic intervention. The symptoms interfere with usual activities of daily living causing discomfort but pose no significant or permanent risk of harm to the study subject.
     * Severe (Grade 3): Events interrupt usual activities of daily living, or significantly effect clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating.

Exclusion Criteria

1. Positive urine pregnancy test at screening or females who intend to become pregnant during the study.
2. COVID-19 signs associated with severe respiratory distress or imminent serious medical outcomes.^^

   ^^Potential Study Subjects Presenting with any of the following should be referred for immediate medical care and are not eligible for the study
   * Fever > 104° F
   * Cough with sputum production
   * Rales and/or rhonchi
   * Difficulty breathing with respiratory distress defined by a respiratory rate ≥30 per minute, heart rate ≥125 per minute, SpO2 ≤93% on room air at sea level or PaO2/FiO2 <300.
   * Persistent pain or pressure in the chest
   * Confusion
3. Any medical disease or condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.
4. Reports a recent positive test result (within the past 6 months) for hepatitis A, hepatitis B or, hepatitis C virus antibody, or HIV-1 antibodies at screening.
5. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 1 month of Study Day 1.
6. Currently enrolled in or plans to participate in another clinical trial with a therapeutic investigational agent (e.g., monoclonal antibody, oral protease inhibitor) that will be received during the study period.
7. History of systemic antiviral therapies (e.g., remdesivir) within the past 30 days.
8. History of oral or parenteral corticosteroid use within the past 30 days. Active use of nasal or inhalable steroids is also exclusionary. Topical steroids are not exclusionary.
9. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to sun exposure.
10. Currently undergoing photodynamic therapy (PDT) or photochemotherapy (PUVA) for an unrelated disease or condition that utilizes photosensitizing drugs including but not limited to 5-aminolevulinic acid, Methyl-5-aminolevulinic acid, porfimer sodium, methoxsalen (8-methoxypsoralen), 5-methoxypsoralen, trioxsalen.
11. Has any oral abnormality (e.g., ulcer, oral candidiasis, oral mucositis, gingivitis) that in the opinion of the investigator would interfere with device use and evaluation.
12. Any intra-oral body piercings that cannot be removed and remain removed for the duration of the study. Metal orthodontia is permitted as braces will be covered by the device mouthpiece.
13. Any individual without teeth or with a dental malformation that precludes directed use of the device as intended.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — EmitBio
Locations (9):
- United States (9):
  - Site 2 - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Site 1 - APF Research LLC, Miami, Florida
  - Site 8 - WellNow Urgent Care, Kalamazoo, Michigan
  - Site 9 - Revival Research Institute, LLC, Sterling Heights, Michigan
  - Site 4 - Peters Medical Research, High Point, North Carolina
  - Site 7 - WellNow Urgent Care, Cincinnati, Ohio
  - Site 5 - WellNow Urgent Care, Columbus, Ohio
  - Site 6 - WellNow Urgent Care, Dayton, Ohio
  - Site 3 - J&S Studies, Inc., College Station, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RD-X19 Device, Dose A: Investigational device that delivers 24 J/cm2
- RD-X19 Device, Dose B: Investigational device that delivers 32 J/cm2
Period: Overall Study
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Started | 28 | 117 | 71
Completed | 26 | 114 | 69
Not Completed | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- RD-X19 Device, Dose A; RD-X19 Device, Dose B: RD-X19. Investigational device that uses safe electromagnetic energy to target the oropharynx.
  RD-X19: Investigational device that uses safe electromagnetic energy to target the oropharynx.
- Total: Total of all reporting groups
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device | Total
Number analyzed (Participants) | 28 | 117 | 71 | 216
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age in years | 38.3 (11.76) | 38.3 (12.57) | 38.6 (13.39) | 38.4 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 63 | 35 | 111
  Male | 15 | 54 | 36 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 24 | 22 | 67
  Not Hispanic or Latino | 7 | 93 | 49 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 18 | 5 | 23
  White | 27 | 94 | 63 | 184
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 28 | 117 | 71 | 216
COVID-19 Composite Severity Score [Mean (Standard Deviation); unit: units on a scale] — Eight symptoms (cough, sore throat, nasal congestion, headache, chills and or sweats, myalgia, fatigue, and nausea (with or without vomiting)) will be rated on a 4-point scale from none (0) to severe (3). The COVID-19 Composite Severity Score is defined as the sum of the eight individual COVID-19 signs and symptoms severity scores divided by eight. Subjects with scores missing for one or more symptoms will have CSS calculated as the sum of all scores reported divided by the number of scores reported
  units on a scale | 1.496 (0.4481) | 1.480 (0.4563) | 1.438 (0.4914) | 1.468 (0.4654)
Baseline disease Severity [Count of Participants; unit: Participants] — Mild COVID-19 • Positive SARS-CoV-2 diagnostic test, viral symptoms, No shortness of breath, dyspnea, abnormal chest imaging, or any other clinical signs indicative of Moderate or Severe COVID-19
  Moderate COVID-19
  • Above with clinical signs suggestive of lower airway involvement, such as resting respiratory rate ≥20 breaths per minute or imaging indicating lower airway disease heart rate ≥ 100 beats per minute, with or an oxygen saturation (SpO2) < 96% but ≥94% on room air at sea level.
  Participants
    Mild COVID | 26 | 64 | 45 | 135
    Moderate COVID | 2 | 53 | 26 | 81

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Resolution of COVID-19 Signs and Symptoms in All Subjects (With Mild or Moderate Disease at Baseline).
Description: Each of eight symptoms (cough, sore throat, nasal congestion, headache, chills and or sweats, myalgia, fatigue, and nausea (with or without vomiting)) will be rated on a 4-point scale from none (0) to severe (3). Time to sustained resolution of COVID-19 signs and symptoms as measured by the time (in hours) when all eight symptoms have been assessed by the subject as none (0) or mild (1) and all symptoms remain at or below 1 until study Day 14. Subjects reporting a persistent fever (100.5 degrees for 36 hours or more) and/or SpO2 levels <96% with any shortness of breath are considered not to have met the success criterion on that day even if all other symptoms are reported as none (0) or mild (1).
Time Frame: Baseline thru Day 14
Population: Cohort B, subjects with mild or moderate disease at baseline. Primary analysis was not performed on Cohort A
Measure: Median (95% Confidence Interval); unit: Time in hours
Groups:
- RD-X19 Device, Cohort A: Investigational Device that delivers 16 J/cm2
Arm/Group | RD-X19 Device, Dose B | RD-X19 Device, Cohort A | Sham Device
Number analyzed (Participants) | 117 | 28 | 57
Time in hours
  Median of Time to Sustained Resolution | 113.5 [99.3 to 142.5] | 172.1 [115.5 to 223.5] | 115.1 [81.9 to 166.3]
  25th Percentile of Time to Sustained Resolution | 63.8 [52.7 to 82.7] | 91.6 [66.0 to 160.7] | 55.4 [42.7 to 81.9]
  75th Percentile of Time to Sustained Resolution | 190.6 [164.5 to 246.3] | 266.3 [192.1 to 384] | 196.6 [166.3 to 294.9]
Statistical Analysis 1: Comparison: RD-X19 Device, Dose B vs Sham Device; Log Rank Test and Cox PH Regression analyses were performed unstratified; Test type: Superiority; p = 0.9784, Regression, Cox; Hazard Ratio (HR) = 1.005, 95% CI 2-sided [0.717 to 1.408]

2. Primary Outcome: Sustained Resolution of COVID-19 Signs and Symptoms in Subjects With Mild Disease at Baseline.
Description: as for outcome 1
Time Frame: Baseline thru Day 14
Population: Cohort B, subject of subjects with mild disease at baseline
Measure: Median (95% Confidence Interval); unit: Time in hours
Groups:
- RD-X19 Device Cohort A: Investigational device that delivers 16 J/cm2
Arm/Group | RD-X19 Device, Dose B | Sham Device | RD-X19 Device Cohort A
Number analyzed (Participants) | 64 | 34 | 26
Time in hours
  Median Time of Sustained Resolution | 99.3 [72.2 to 119.3] | 119.5 [78.0 to 185.6] | 172.1 [101.8 to 223.5]
  25th Percentile of Time to Sustained Resolution | 54.8 [45.1 to 72.2] | 47.9 [42.7 to 93.0] | 87.9 [66.0 to 160.7]
  75th Percentile of Time to Sustained Resolution | 164.8 [120.3 to 222.3] | 196.6 [144.0 to 322.0] | 254.7 [192.1 to 384]
Statistical Analysis 1: Comparison: RD-X19 Device, Dose B vs Sham Device; Test type: Superiority; p = 0.1512, Regression, Cox — Log Rank Test and Cox PH Regression analyses were performed unstratified; Hazard Ratio (HR) = 1.388, 95% CI 2-sided [0.887 to 2.172]

3. Secondary Outcome: Medically Attended Visits
Description: Numbers and percentages of study subjects who require medical attention or intervention attributed to COVID-19;
Time Frame: Baseline thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 5 | 5 | 2

4. Secondary Outcome: Severe Disease Progression
Description: Numbers and percentages of study subjects who progress to severe disease with respiratory rate >30/minute and/or O2 saturation </=93% on room air or FiO2 ≥300% with any respiratory distress.
Time Frame: Baseline thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 3 | 2 | 1

5. Secondary Outcome: Hospitalizations
Description: Numbers and percentages of study subjects who require hospitalization for severe COVID-19.
Time Frame: Baseline thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 4 | 3 | 2

6. Secondary Outcome: Worsening of Disease
Description: Number and percentage of study subjects who experience progression of COVID-19 as defined by an increase of the composite COVID-19 severity score greater than baseline at any point in the study on or after day 3.
Time Frame: Day 3 thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 5 | 10 | 11

7. Secondary Outcome: Return to Pre-COVID Health
Description: Numbers and percentages of study subjects on day 8 and day 14 who answer yes to the following patient-reported global impression assessments, a) return to usual health and b) return to usual activities.
  1. In the past 24 hours, have you returned to your usual health (before your COVID-19 illness)? Yes or No
  2. In the past 24 hours, have you returned to your usual activities (before your COVID-19 illness)? Yes or No
  Note: subjects with missing Data at Day 8 or Day 14 were not included in total subjects analyzed
Time Frame: Days 8 and 14
Population: Visit 4/Day8
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants
  Subjects who returned to usual health on Day 8 | 10 | 54 | 27
  Subjects who returned to usual activities on Day 8 | 9 | 74 | 41
  Subjects who returned to usual health on Day 14: number analyzed (Participants) | 27 | 114 | 69
  Subjects who returned to usual health on Day 14 | 17 | 84 | 49
  Subjects who returned to usual activities on Day 14: number analyzed (Participants) | 27 | 114 | 69
  Subjects who returned to usual activities on Day 14 | 16 | 96 | 56

8. Secondary Outcome: Mean Change in Nasopharyngeal Viral Load
Description: Mean change in nasopharyngeal viral load from baseline on days 3, 5, 8, and 14.
Time Frame: Days 3, 5, 8 and 14
Population: Subjects with Mild and Moderate Disease at Baseline
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 22 | 114 | 67
Log10 copies/mL
  Day 3 | -0.849 (0.8828) | -1.269 (1.0666) | -0.928 (1.7048)
  Day 5 | -2.218 (0.9273) | -2.649 (1.6975) | -2.107 (1.9003)
  Day 8 | -3.663 (1.8057) | -4.132 (1.9791) | -3.744 (1.8545)
  Day 14 | -4.827 (1.6769) | -5.584 (1.5876) | -5.084 (2.1024)

9. Secondary Outcome: Proportion of Subjects Demonstrating Clearance of Viral Infection
Description: Proportion of subjects demonstrating clearance of viral infection on Days 3, 5, 8 and 14.
Time Frame: Days 3, 5, 8 and 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 22 | 114 | 67
Participants
  Day 3 | 0 | 2 | 4
  Day 5 | 0 | 15 | 6
  Day 8 | 1 | 34 | 19
  Day 14 | 2 | 68 | 34

10. Secondary Outcome: Day 8 Composite Resolution
Description: Proportion of study subjects who achieve Day 8 Composite Resolution.
Time Frame: Baseline thru Day 8
Population: N (%) subjects achieving success on Composite Resolution
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 25 | 113 | 70
Participants | 14 | 81 | 48

11. Secondary Outcome: Endotracheal Ventilation or ECMO
Description: Number and percentage of study subjects who require endotracheal ventilation or ECMO with or without the use of solumedrol.
Time Frame: Baseline thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 0 | 0 | 0

12. Secondary Outcome: Death
Description: Number and percentage of study subjects who die.
Time Frame: Baseline thru Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
Number analyzed (Participants) | 28 | 117 | 71
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through day 14 (±2 days)
Arm/Group | RD-X19 Device, Dose A | RD-X19 Device, Dose B | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/117 | 0/71
Serious Adverse Events (participants affected / at risk) | 4/28 | 3/117 | 2/71
Other Adverse Events (participants affected / at risk) | 19/28 | 55/117 | 39/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD-X19 Device, Dose A (N=28) | RD-X19 Device, Dose B (N=117) | Sham Device (N=71)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RD-X19 Device, Dose A (N=28) | RD-X19 Device, Dose B (N=117) | Sham Device (N=71)
Administrative Site Pain (General disorders) | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 3 | 13 | 11
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 2 | 6 | 7
Fatigue (General disorders) | 1 | 11 | 6
Malaise (General disorders) | 1 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 4 | 5 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0
Neutrophil/Lymphocyte Ratio Increased (Investigations) | 1 | 7 | 4
Red Cell Distribution Width Increased (Investigations) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Jaw Clicking (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 10
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data and reports of study data are the property of the study sponsor. The sponsor may grant the PI the right to publish the results of this research in a scientific journal, conditional upon the review and concurrence of the sponsor

DOCUMENTS (2):
  • Study Protocol (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04966013/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04966013/SAP_001.pdf